CLINICAL TRIAL: NCT07034287
Title: eGAPcare: Modifying the Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention in the Emergency Department for Telehealth
Brief Title: Modifying the Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention in the Emergency Department for Telehealth
Acronym: eGAPcare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-1370
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Older Adults (65 Years and Older); Fall Prevention; Telehealth; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Telehealth physical therapy and pharmacy consultation at baseline emergency department visit.
  Interventions: Other: Telehealth physical therapy and pharmacy consultation

INTERVENTIONS:
Other: Telehealth physical therapy and pharmacy consultation — Telehealth physical therapy and pharmacy consultation at baseline emergency department visit.

SUMMARY:
The goal of this clinical trial is to determine the feasibility of eGAPcare, a telehealth modification of the GAPcare fall prevention intervention, in older adults in a community emergency department. The main questions it aims to answer are:

* Can telehealth physical therapy and pharmacy consultations be conducted in a community emergency department?
* Does the telehealth modification of GAPcare decrease recurrent falls at 6 months? Participants will
* Receive telehealth physical therapy and pharmacy consultation while in the emergency department
* Participate in follow-up visits over the phone for 6 months following the initial emergency department visit
* Complete study questionnaires delivered by study staff.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adult (non-institutionalized) 65 years-old or older presenting to ED after a fall
* Fall not due to syncope or external force (i.e., struck by car or assault)
* Fall not due to serious illness (i.e., stroke, acute myocardial infarction)
* Will be discharged to home/assisted living/rehabilitation at completion of ED visit (i.e., not admitted)
* Proxy available to give informed consent if patient lacks capacity

Exclusion Criteria:

* Unable to give informed consent due to intoxication or acute change in mental status
* Presence of injuries that prevent mobilization (i.e., pelvic or lower extremity fractures)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported or caregiver reported falls | Within 6 months of the initial emergency department visit
Electronic Health Record reported falls and healthcare usage | Within 6 months of the initial emergency department visit

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No